CLINICAL TRIAL: NCT03073434
Title: Pregnancy Outcomes in Renal Transplant Recipients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 15-289
Record Dates: First submitted 2017-02-13; First posted 2017-03-08 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Renal Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective study involving all patients with a history of renal transplant that attended antenatal clinics at various Toronto hospitals and subsequently delivered between January 2000 and December 2014.

The purpose of this study is to describe the incidence of adverse pregnancy-and transplant-related outcomes, and report placental ultrasound and placental pathology findings in renal transplant recipients with contemporary standards of care in Toronto.

This study also seeks to determine whether factors such as maternal age, transplant-to-pregnancy interval, hypertension, diabetes mellitus, treatment regimens, and the primary cause for renal failure are associated with higher risk of adverse pregnancy outcomes in renal transplant recipients.

DETAILED DESCRIPTION:
Adverse pregnancy outcomes in women with renal transplants have been attributed to a number of factors. A recent systematic review suggested an association between maternal age and adverse pregnancy outcomes such as miscarriage and stillbirth. There are also some data to suggest that maternal hypertension, diabetes mellitus, elevated serum creatinine and proteinuria and some medications such as cyclosporine are associated with adverse pregnancy outcomes such as preeclampsia, intrauterine growth restriction and preterm delivery.There is no consensus on whether the transplant-to-pregnancy interval is associated with adverse pregnancy outcomes. As well, it is not clear if the findings of other studies will also hold true in a Toronto population.

This study seeks to answer the following questions:

1. What is the incidence of adverse transplant- and pregnancy-related adverse outcomes in renal transplant recipients that have had pregnancies between 2000 and 2014 in Toronto and how does this compare with earlier data from Toronto and with recently published data?
2. Are factors such as maternal age, transplant-to-pregnancy interval, hypertension, diabetes mellitus, specific treatment regimens and the primary cause for renal failure associated with an increased risk of adverse pregnancy- and transplant-related adverse outcomes in these women?

ELIGIBILITY:
Inclusion Criteria:

* All patients with a history of renal transplant that attended antenatal clinics at Mt. Sinai Hospital, Sunnybrook Health Sciences Centre and St. Michael's hospital and subsequently delivered between January 2000 and December 2014

Exclusion Criteria:

* Patients who do not meet the above criteria are excluded from the sample

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: All patients with a history of renal transplant that attended antenatal clinics at Mt. Sinai Hospital, Sunnybrook Health Sciences Centre and St.Michael's hospital and subsequently delivered between January 2000 and December 2014.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Maternal health outcomes obtained from patient medical record | From start of pregnancy (1 week gestation) to 6 weeks post-partum
  Observed health outcomes of the mother after giving birth, obtained retrospectively from the patient's medical record.
Fetal and neo-natal health outcomes obtained from patient medical record | From start of pregnancy (1 week gestation) to 6 weeks post-partum
  Observed health outcomes of the fetus/neonate after delivery, obtained retrospectively from the patient's medical record.
Placental outcomes obtained from patient medical record | Measured immediately after delivery
  Biochemistry and physical characteristics of the placenta, obtained retrospectively from the patient's medical record.
Transplant-related outcomes obtained from patient medical record | From start of pregnancy (1 week gestation) to 6 weeks post-partum
  Graft function during pregnancy and at end of pregnancy, obtained retrospectively from the patient's medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Berger, MD, Principal Investigator — Unity Health Toronto

IPD SHARING:
Plan to Share IPD: No